CLINICAL TRIAL: NCT05614518
Title: A Randomized, Open-Label, Crossover, Controlled, Multi-center Clinical Study to Assess the Diagnostic Performance and Safety of 18F-NaF-PET/CT in Bone Metastases of Malignant Tumors Compared With 99mTc⁃MDP-BS±SPECT
Brief Title: Diagnostic Performance and Safety of 18F-NaF-PET/CT in Bone Metastases Compared With 99mTc⁃MDP-BS±SPECT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: HTA Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: BJK-Z-F18HN-202010-YZGK
Record Dates: First submitted 2022-10-30; First posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Bone Metastases
Keywords: Lung Cancer; Breast Cancer; Prostate Cancer
MeSH Terms: conditions — Lung Neoplasms; Breast Neoplasms; Prostatic Neoplasms | interventions — Technetium Tc 99m Medronate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 18F-NaF-PET/CT (Experimental): Patients undergo an 18F-NaF-PET/CT scan and an 99mTc-MDP-BS±SPECT scan within a time frame of 7 days.
  Generic Name: Sodium Fluoride F-18 injection Dosage Form: Injection Dosage: Administer 5-10 mCi as an intravenous injection Frequency and Duration: Single dose
  Interventions: Drug: Sodium Fluoride F-18 Injection
- 99mTc-MDP-BS±SPECT (Active Comparator): Patients undergo an 18F-NaF-PET/CT scan and an 99mTc-MDP-BS±SPECT scan within a time frame of 7 days.
  Generic Name: Technetium[99mTc] Methylenediphosphonate Injection Dosage Form: Injection Dosage: Administer 10-25 mCi as an intravenous injection Frequency and Duration: Single dose
  Interventions: Drug: Technetium[99mTc] Methylenediphosphonate Injection

INTERVENTIONS:
Drug: Sodium Fluoride F-18 Injection — Each subject was given 5-10 mCi intravenously. Images were collected 90-120 min after injection.
  Other Names: 18F-NaF Injection
  Arms: 18F-NaF-PET/CT
Drug: Technetium[99mTc] Methylenediphosphonate Injection — Each subject was given 10-25 mCi intravenously. Images were collected 3-6 hours after injection.
  Other Names: 99mTc-MDP Injection
  Arms: 99mTc-MDP-BS±SPECT

SUMMARY:
The goal of this clinical trial was to assess the diagnostic performance and safety of Sodium Fluoride F-18 Positron Emission Tomography / Computed Tomography (18F-NaF-PET/CT) in bone metastases of malignant tumors compared with Technetium[99mTc] Methylenediphosphonate Bone Scintigraphy ± Single Photon Emission Computed Tomography (99mTc-MDP-BS±SPECT).

The enrolled subjects were randomly assigned to two sequences A and B at a ratio of 1:1. Within 7 days, 18F-NaF-PET/CT and 99mTc-MDP-BS±SPECT bone imaging were performed alternately.

The sensitivity, specificity, positive and negative predictive value of 18F-NaF-PET/CT and 99mTc-MDP-BS±SPECT were calculated respectively based on the diagnostic data of standard of truth.

ELIGIBILITY:
1. Male or female, age 18 to 75 years, inclusive.
2. It is confirmed to be lung cancer, prostate cancer or breast cancer by combining medical history, imaging and pathological examination, and radionuclide bone imaging is required, and any one of the following is required:

   1. Bone imaging within 3 months before the signing the ICF cannot exclude bone metastasis.
   2. Associated with clinical manifestations related to bone metastasis, including bone pain, activity disorder, pathological fracture, spinal cord or spinal nerve compression symptoms, alkaline phosphatase elevation, hypercalcemia or Prostate Specific Antigen (PSA) >10 ng / ml.
   3. Those with definite metastasis outside the primary tumor focus.
   4. Patients with a history of bone metastasis.
   5. Patients who need to confirm the status of bone metastasis for tumor staging.
3. According to the standard of the Eastern Cooperative Oncology Group (ECOG), the score was 0-1.
4. The expected survival of the Patients was > 6 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2022-06-02 (Actual); Study Completion 2022-06-02 (Actual)

PRIMARY OUTCOMES:
Assess the sensitivity and specificity of 18F-NaF-PET/CT compared with 99mTc-MDP-BS±SPECT based on subjects. | After the completion of two scanning imaging (or extended to 6 months).
  The sensitivity and specificity of 18F-NaF-PET/CT and 99mTc-MDP-BS±SPECT were calculated respectively based on subjects according to Standard of Truth.

SECONDARY OUTCOMES:
Number of participants with adverse events as assessed by CTCAE v5.0. | From the first day of administration to the end of the trial.
  Any adverse events were recorded from the first day of administration to the end of the trial. Adverse events were assessed by CTCAE v5.0.
Assess the positive and negative predictive value of 18F-NaF-PET/CT compared with 99mTc-MDP-BS±SPECT based on subjects. | After the completion of two scanning imaging (or extended to 6 months).
  The positive and negative predictive value of 18F-NaF-PET/CT and 99mTc-MDP-BS±SPECT were calculated respectively based on the diagnostic data of Standard of Truth.
Assess the sensitivity, specificity, positive and negative predictive value of 18F-NaF-PET/CT compared with 99mTc⁃MDP-BS±SPECT based on lesions. | After the completion of two scanning imaging (or extended to 6 months).
  The sensitivity and specificity of 18F-NaF-PET/CT and 99mTc-MDP-BS±SPECT were calculated respectively based on lesions according to Standard of Truth.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Academy of Medical Sciences Peking Union Medical College Hospital, Beijing, China